CLINICAL TRIAL: NCT04071860
Title: Developing a Non-contact Sleep Apnoea Detector, Suitable for Home Studies- The Safescan Study.
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Iceni Labs Ltd, Warwickshire, United Kingdom (Unknown)
Responsible Party: Sponsor
Other Study IDs: P02423
Record Dates: First submitted 2019-03-04; First posted 2019-08-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Sleep Apnoea; Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- discovery and learning cohort: Data from this cohort will be used to develop the software algorithms
- Validation: Data from this cohort will be used to validate the software algorithms

SUMMARY:
Sleep apnoea (SA) is a common condition in adults and children that causes disturbed sleep and daytime symptoms. It is characterised by disrupted breathing with disturbed sleep patterns. In adults this can lead to dangerous daytime sleepiness affecting for example driving performance. In children it may lead to hyperactivity in the day and poor school performance. There are a number of techniques for diagnosing the disorder but they can affect the quality of sleep which sometimes makes them inaccurate. Most are unsuitable for small children who cannot understand the value of the tests and tend to remove the monitoring wires and devices in the night. This study aims to validate a new non contact device "Safescan", based on low power radar technology, which can be put under a bed and record breathing patterns with no measuring device in contact with the sleeper. In this initial study the device will be validated in adults, against the gold standard of polysomnography (PSG) in the sleep laboratory at Royal Papworth Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to give informed consent

Exclusion Criteria:

* Patient with known sleep disordered breathing using a treatment device (e.g. continuous positive airway pressure) on the night of the study.
* Polysomnography study records less than 4 hours of respiratory data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the sleep laboratory for inpatient polysomnography, irrespective of working or known diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Agreement between the Apnoea hypopnea index (AHI) per hour as measured overnight by the Safescan device and by clinical polysomnography | overnight (8-10 hours)
  Agreement in AHI +/- 10% between Safescan device and PSG. A comparison will be made between the 2 AHI's for each participant. The proportion in whom there is an agreement within +/- 10% will be reported.

SECONDARY OUTCOMES:
Agreement between the Safescan device respiratory rate (RR) as breaths per minute overnight and RR from PSG | overnight (8-10 hours)
  Agreement +/- 1 breath per minute between Safescan device and PSG
Agreement in recorded body position between Safescan device and PSG | overnight (8-10 hours)
  Percentage of 1 minute epochs during the the Safescan body position is in agreement with that of the PSG

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, MD, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No